CLINICAL TRIAL: NCT05952388
Title: Impact of Clinical Pharmacy Services on Medication Cost and Hospitalization Rates in Hemodialysis Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left the institution & this is not an applicable clinical trial (ACT).
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HRRC # 02-423
Record Dates: First submitted 2008-07-09; First posted 2023-07-19 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: End Stage Renal Disease
Keywords: Document the number, type, and severity of DRPs; in HD patients.; Determine the rates and categorization of; DRPs-associated hospitalizations in HD patients.; Document the number and types of pharmaceutical; Care Interventions.; Determine the outcomes of pharmaceutical care; Intervention; Determine the rate of acceptance of pharmaceutical; Care Interventions .; Assign significance rank to pharmaceutical; Determine annual drug cost in HD patients.; Determine drug cost associated for treatment; of each HD patient comorbidity.; Determine Quality of Life (QoL) using a renal; -specific instrument
MeSH Terms: conditions — Kidney Failure, Chronic; Limb-girdle muscular dystrophy, type 2C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Behavioral Patient Care (No Intervention): Chart review
  Interventions: Other: Behavioral Patient care

INTERVENTIONS:
Other: Behavioral Patient care — chart review
  Other Names: Chart review

SUMMARY:
The purpose of this study is to evaluate the effects of pharmaceutical care interventions in the ambulatory hemodialysis patients over a one-year period. Cost containment occurs through pharmaceutical care interventions designed to identify and ameliorate drug-related problems (DRPs), improve the cost-effectiveness of therapeutic regimens and prevent hospitalizations.

DETAILED DESCRIPTION:
Approximately 350,000 end-stage renal disease (ESRD) patients in the United States utilized over $17.9 billion Medicare dollars in 1999. The ESRD population and cost is projected to double by 2010. ESRD patients have a mean of 5 comorbidities per patient and are prescribed a median of eight medications. The average monthly medication cost per patient is approximately $1,200.00. For every dollar spent on medication an additional $1.77 is spent on drug-related problems (DRPs). Dialysis patients are at high risk for DRPs. It is unknown if continued pharmacist intervention in hemodialysis patients will improve patient care, reduce medication utilization and cost, and prevent hospitalization as seen in other populations. The purpose of this study is to investigate the impact of continued pharmacist intervention in ambulatory hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible for inclusion in the study if they have been on HD for greater than three months, greater than 18 years of age, those who plan to be continuously enrollment in therapy at the same dialysis center throughout the duration of the study. Informed consent will be obtained on eligible patients. The study is to be approved by the Human Research Review Committee prior to initiation.

Exclusion Criteria:

* Patients will be excluded if they have been on HD for less than three months, decline the opportunity to participate, or are less than 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2003-01 (Actual); Primary Completion 2003-01 (Actual); Study Completion 2003-01 (Actual)

PRIMARY OUTCOMES:
Reduction in at home medications | through study completion, an average of 1 year
  Behavioral: Patent care

CONTACTS AND LOCATIONS:
Overall Officials: Amy B Pai, Pharm.D, Principal Investigator — University of New Mexico